CLINICAL TRIAL: NCT05720702
Title: A Feasibility Trial of One-carbon Metabolism Cofactor Supplements for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Feasibility Trial of OCM Supplements for the Treatment of NAFLD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112107
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Homocysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAFLD Group (Experimental): The NAFLD group will be asked to take Hcy lowering supplements (Vitamin B12, Folate, Vitamin B6, and Betaine) daily for 12 weeks. Over the course of approximately 12 to 13 weeks, participants will complete two in person visits and two phone visits. During the in person visits NAFLD participants will complete the following activities:
  Review medical history; Physical examination; Vital signs (blood pressure, heart rate, respiratory rate, body temperature); Measure height, weight, body mass index, and waist circumference; Grip test; Fasting blood tests; Pregnancy test (if applicable); Fibroscan with CAP score; QOL questionnaire
  Interventions: Dietary Supplement: homocysteine (Hcy) lowering supplements

INTERVENTIONS:
Dietary Supplement: homocysteine (Hcy) lowering supplements — NAFLD participants will take homocysteine (Hcy) lowering supplements daily for 12 weeks.

SUMMARY:
The purpose of the study is to assess the feasibility of a trial to test the effects of homocysteine (Hcy) lowering supplements in patients with NAFLD.

NAFLD patients will be asked to take Hcy lowering supplements (Vitamin B12, Folate, Vitamin B6, and Betaine) daily for 12 weeks. Over the course of approximately 12 to 13 weeks, participants will complete two in person visits and two phone visits to complete activities such as physical exam, fibroscan, blood draws, and questionnaires.

DETAILED DESCRIPTION:
The purpose of the study is to assess the feasibility of a trial to test the effects of homocysteine (Hcy) lowering supplements in patients with NAFLD.

NAFLD patients will be asked to take Hcy lowering supplements (Vitamin B12, Folate, Vitamin B6, and Betaine) daily for 12 weeks. Over the course of approximately 12 to 13 weeks, participants will complete two in person visits and two phone visits. During the in person visits NAFLD participants will complete the following activities:

* Review medical history
* Physical examination
* Vital signs (blood pressure, heart rate, respiratory rate, body temperature)
* Measure height, weight, body mass index, and waist circumference
* Grip test
* Fasting blood tests
* Pregnancy test (if applicable)
* Fibroscan with CAP score
* QOL questionnaire

ELIGIBILITY:
We will enroll NAFLD patients, blocked by age 50 years (≤ 50; > 50) and sex (M; F, four patients/subjects in each block).

Inclusion Criteria for NAFLD Group:

1. Increased hepatic fat accumulation diagnosed by either abdominal ultrasound or CT AND elevated CAP score of 280 dB/m or higher
2. HOMA-IR ≥ 2 or the diagnosis of metabolic syndrome
3. Chronic elevation of transaminases: ALT elevation (more than 2 times during the past 12 months, defined by 19 U/L for women and 30 U/L for men 31)
4. Stable use of any potential anti-NASH therapy (i.e., vitamin E, pioglitazone, glucagon like peptide 1 agonist, etc.) for 6 months prior to screening.
5. Aged 18+ years
6. Able to provide legal consent

Exclusion Criteria for NAFLD Group:

1. Any contraindication to the study supplements
2. Inability to obtain valid fibroscan measures at the screening
3. Pregnancy or lactation
4. Clinical diagnosis of cirrhosis or other chronic liver diseases
5. Recent use of steatogenic medications
6. Excess alcohol use (>21/ >14 drinks weekly in men/women)
7. Chronic kidney disease
8. Supplement use within 30 days, containing any of the study supplements
9. Total parenteral nutrition
10. Any clinical conditions associated with malabsorption
11. Any active diagnosis of malignancy
12. Use of immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
FibroScan-aspartate aminotransferase (FAST) score | 12 weeks
  To minimize interindividual variability of fibroscan measurements, all of the fibroscan will be performed by a single, experienced operator using the same probe (M vs. XL) and technique for the paired measurements. The FibroScan-aspartate aminotransferase (FAST) score is a simple algorithm that can diagnose NASH using an elevated (≥ 4) NAFLD activity score (NAS) and significant fibrosis score (≥ 2).

SECONDARY OUTCOMES:
Feasibility as measured by percentage of completion of enrollment | 4 months
  The trial design will be considered feasible if at least 13 NAFLD patients (≥80%) are enrolled over the 4-month period
Assess safety of the trial. | 12 weeks
  Based on reported adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Ayako Suzuki, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to share IDP with other researchers at this time.